CLINICAL TRIAL: NCT05001087
Title: A "Physician & Patient-powered" Cohort Registry
Brief Title: A "Physician & Patient-powered" Cohort Registry (MY MYELOMA)
Acronym: MY MYELOMA
Status: Recruiting | Type: Observational
Sponsor: Fondazione EMN Italy Onlus (Other)
Collaborators: Amgen (Industry); GlaxoSmithKline (Industry); Janssen-Cilag S.p.A. (Industry); Sanofi (Industry); Takeda (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: 535/2020
Record Dates: First submitted 2021-01-22; First posted 2021-08-11 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients registry: Non-interventional, multicentre, retrospective and prospective registry. In order to increase the sample size and the validity of the Registry, patients who were diagnosed with myeloma since 1st January 2019 will also be included retrospectively, once their informed consent has been obtained by the enrolling centre. Being a registry, patients will be enrolled consecutively according to their appointments at the centre, at the discretion of their doctor and only once the patient has signed the informed consent form.
  Also patients participating in interventional or other observational studies can be enrolled. In case of patients enrolled in interventional trials, only baseline and survival data can be collected for the period in with the patient is in interventional trial.
  The data will be collected using an electronic data capture (EDC) platform. Hospital visits are planned every 6 months.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Not applicable-Observational study

SUMMARY:
The aim of this observational study is the creation of a national multiple myeloma registry to monitor the current routine clinical practice in Italy and describe the standard of care adopted for the diagnosis and treatment of patients with multiple myeloma in the different Italian hematology centers.

DETAILED DESCRIPTION:
In Italy, myeloma accounts for 1.3% of all tumour diagnoses in males and for 1.2% of all tumour diagnoses in women. The incidence is 9.5 new cases per 100,000 males and 8.1 cases per 100,000 females. Median age at diagnosis is 68 years and approximately 2% of patients experience onset before the age of 4011. Therefore is to establish a national disease registry to monitor current routine clinical practice in Italy and to describe the standard of care adopted for the diagnosis and treatment of patients with myeloma. National registries have already been established in some countries and a recently-published meta-analysis highlighted certain differences in treatment, survival and the demographic characteristics of patients. An Italian national registry is important for analysing the current situation, in order to deal with the changes that lie ahead. In addition to the standard epidemiological registry - as described in the statistical methods section - a patientpowered registry (PPR) will also be established to encourage patient participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* Age ≥ 18 years
* Diagnosis of active/symptomatic multiple myeloma (according to CRAB and biological parameters) no earlier than 1st January 2019
* Able and willing to sign an informed consent form

Exclusion Criteria:

* None considered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will include approximately 30 Italian haematology facilities. On the basis of the centres' enrolment capacity and incidence and epidemiology data it is reasonable to presume that at least 1900 patients will be enrolled in 3 years. Only patients who meet the eligibility criteria will be included in the registry.
Sampling Method: Probability Sample
Enrollment: 1900 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 3 years
  Time between diagnosis and death.
Time to next treatment (TTNT) | 3 years
  Time to next treatment will be measured from the screening to the date of next anti-myeloma therapy, for each treatment regime.

SECONDARY OUTCOMES:
Patient reported outcomes (PROs) | 3 years
  Periodic completion of the EORTC-QLQ-C30 to evaluate the quality of life of the patients.
Costs incurred by the patients | 3 years
  Evaluation of the costs incurred by the patients related to the therapy based on the different treatments.

CONTACTS AND LOCATIONS:
Locations (27):
- Italy (27):
  - A.O.U di Careggi, Florence, Firenze
  - AOU Ospedali Riuniti Umberto I, Ancona
  - Policlinico di Bari - Ematologia con Trapianto, Bari
  - Policlinico di Bari, Bari
  - Policlinico S. Orsola, Bologna
  - A.O. Spedali Civili di Brescia, Brescia
  - AOU Policlinico Vittorio Emanuele, Catania
  - A.O.U Policlinico S. Martino, Genova
  - ASST Santi Paolo e Carlo, Milan
  - Fondazione IRCCS Ca' Grande Ospedale Maggiore Policlinico, Milan
  - Istituto Nazionale Tumori, Milan
  - Ospedale Niguarda Cà Grande, Milan
  - Ospedale San Gerardo di Monza, Monza
  - A.O.U Federico II, Napoli
  - Ospedale Maggiore, Novara
  - A.O.U di Parma, Parma
  - Policlinico San Matteo Fondazione IRCCS, Pavia
  - Ospedale "Infermi", Rimini
  - Ospedale S. Eugenio, Roma
  - Policlinico Umberto I - Università La Sapienza, Roma
  - Policlinico Universitario Campus Biomedico, Roma
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - A.O. Santa Maria, Terni
  - A.O Ordine Mauriziano, Torino
  - AOU Città della Salute e della Scienza di Torino, Torino
  - Policlinico Universitario di Udine, Udine
  - Ospedale di Circolo, Varese